CLINICAL TRIAL: NCT00651521
Title: Clinical Feature and Outcome of Angiographic Coronary Artery Disease in Chronic Kidney Disease Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, I Wen Wu, MD, Attending physician, Chang Gung Memorial Hospital
Other Study IDs: IWW-0002; CGMH-IRB-96-1680B
Record Dates: First submitted 2008-03-30; First posted 2008-04-02 (Estimated); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Coronary Artery Disease; Chronic Kidney Disease
Keywords: Angiographic CAD; Chronic kidney disease; Left ventricular dysfunction; Body mass index; Cardiovascular mortality; Coronary angiography
MeSH Terms: conditions — Coronary Artery Disease; Renal Insufficiency, Chronic; Ventricular Dysfunction, Left

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (6):
- 1: CKD stage 1 patients
- 2: CKD stage 2 patients
- 3: CKD stage 3a patients
- 4: CKD stage 3b patients
- 5: CKD stage 4 patients
- 6: CKD stage 5 patients

SUMMARY:
The prevalence and mortality rate of cardiovascular disease (CVD) in chronic kidney disease (CKD) patients is high. The prevalence of coronary artery disease (CAD) in CKD population ranges from 38 to 65%, with an average of 3.3 coronary lesions per person. The relative risk for death from myocardial infarction and CAD is 1.18 in CKD patients with GFR < 60 ml/min. Because of this high prevalence of CAD and its high mortality, reducing and preventing CAD risk factors is crucial in the clinical management of CKD patients.

Low glomerular filtration rate (GFR) constitutes an important independent risk factor for CAD. Several pathogenic factors play role in the genesis of cardiovascular dysfunction in chronic kidney disease. Increased traditional CAD risk factor, endothelial dysfunction, sympathetic hyperactivity, renin-angiotensin system activation, increased glycosylated end products, all contribute to the characteristic medial calcification of cardiovascular disease in CKD patients. Hypertension, fluid overloading and anemia further aggravated the cardiac loading, leading to myocardial hypertrophy with chamber dilatation, heart failure and death.

The mortality rate of CAD in CKD patients is extremely high. The NHANES II (National Health and Nutritional Evaluation Survey) found an increased of mortality rate> 51%, when the GFR decreased from > 90 to < 70 ml/min. The 1-year mortality rate in different CKD stage were 0.7% (normal renal function patients), 2.0% (patients with proteinuria), 3.5% (overt proteinuric patients) and 12.1% (dialysis patients), respectively. However, the clinical feature and outcome of CAD in different stage of CKD remains unclear.

We conducted a retrospective cohort study involving all patients admitted for coronary angiography from 1992 to 2004. The patients were categorized into five stages of CAD to compare the risk factor, clinical feature and outcome. Determination of this relationship can help to establish factors for early detection of CAD in CKD patients and also prognostic factor to improve outcome of these patients.

DETAILED DESCRIPTION:
All patients who underwent cardiac catheterization for assessment of CAD at Keelung Chang Gung Memorial Hospital between 1992 and 2004 with continuous serum creatinine values measured before admission were included in this analysis. Data were obtained from medical records of the database center of our institution. Demographic and clinical data were assessed. The age, sex, body mass index (BMI), body surface area (BSA), underlying comorbidities, CAD risk factors (including diabetes mellitus, hypertension, dyslipidemia, smoking, and obesity, defined as a BMI > 30) and clinical presentation were included in this study. Hemodynamic parameters including the systolic and diastolic blood pressure, heart rate and left ventricular ejection fraction were also obtained. Coronary angiography was performed using a low-osmolarity non-ionic contrast medium (iodixanol) by experienced cardiologist. Coronary artery disease was defined as a 50% or greater lumen narrowing of a major epicardial artery or its branches. A left main stenosis of 50% or greater was regarded as equivalent to 2-vessel disease. Blood samples were collected during admission before angiographic procedure. Values of hemoglobin, white blood cells, platelet, high sensitivity C-reactive protein (hs-CRP) and troponin I was included. The treatment modality was divided into three categories: medical, percutaneous coronary intervention (PCI, including balloon angioplasty with or without stent placement) and coronary artery bridge graft (CABG) on the basis of clinical condition and angiographic finding. The outcome was followed-up until 12 months after angiographic procedure. The estimated total study patient number is approximately 1000 patients.

ELIGIBILITY:
Inclusion Criteria:

1. CKD patients with typical angina or positive electrocardiographic finding for myocardia ischemia.
2. Aged 20-80 years.

Exclusion criteria:

1. recipient of renal transplant graft or dialysis therapy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All CKD patients admitted for coronary angiography from 1992 to 2019. The patients were further categorized into five stages of CKD.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2009-04; Primary Completion 2022-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
all cause death | 10 years
  number of death
change of renal function | 10 years
  number to dialysis

CONTACTS AND LOCATIONS:
Overall Officials: Iwen Wu, MD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Department of Nephrology,Chang Gung Memorial Hospital, Keelung, Taiwan

REFERENCES:
- [Background] Aronow WS, Ahn C, Mercando AD, Epstein S. Prevalence of coronary artery disease, complex ventricular arrhythmias, and silent myocardial ischemia and incidence of new coronary events in older persons with chronic renal insufficiency and with normal renal function. Am J Cardiol. 2000 Nov 15;86(10):1142-3, A9. doi: 10.1016/s0002-9149(00)01176-0. PMID 11074216
- [Background] Reddan DN, Szczech L, Bhapkar MV, Moliterno DJ, Califf RM, Ohman EM, Berger PB, Hochman JS, Van de Werf F, Harrington RA, Newby LK. Renal function, concomitant medication use and outcomes following acute coronary syndromes. Nephrol Dial Transplant. 2005 Oct;20(10):2105-12. doi: 10.1093/ndt/gfh981. Epub 2005 Jul 19. PMID 16030030
- [Background] Reddan DN, Szczech LA, Tuttle RH, Shaw LK, Jones RH, Schwab SJ, Smith MS, Califf RM, Mark DB, Owen WF Jr. Chronic kidney disease, mortality, and treatment strategies among patients with clinically significant coronary artery disease. J Am Soc Nephrol. 2003 Sep;14(9):2373-80. doi: 10.1097/01.asn.0000083900.92829.f5. PMID 12937316
- [Background] Reis SE, Olson MB, Fried L, Reeser V, Mankad S, Pepine CJ, Kerensky R, Merz CN, Sharaf BL, Sopko G, Rogers WJ, Holubkov R. Mild renal insufficiency is associated with angiographic coronary artery disease in women. Circulation. 2002 Jun 18;105(24):2826-9. doi: 10.1161/01.cir.0000021597.63026.65. PMID 12070108
- [Background] Stack AG. Coronary artery disease and peripheral vascular disease in chronic kidney disease: an epidemiological perspective. Cardiol Clin. 2005 Aug;23(3):285-98. doi: 10.1016/j.ccl.2005.04.003. PMID 16084278
- [Background] Keough-Ryan TM, Kiberd BA, Dipchand CS, Cox JL, Rose CL, Thompson KJ, Clase CM. Outcomes of acute coronary syndrome in a large Canadian cohort: impact of chronic renal insufficiency, cardiac interventions, and anemia. Am J Kidney Dis. 2005 Nov;46(5):845-55. doi: 10.1053/j.ajkd.2005.07.043. PMID 16253724